CLINICAL TRIAL: NCT00090389
Title: New England School of Acupuncture (NESA) Acupuncture Research Collaborative
Brief Title: Acupuncture for Women's Health Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U19AT002022 (NIH)
Record Dates: First submitted 2004-08-25; First posted 2004-08-26 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Ovarian Neoplasms; Endometriosis; Pelvic Pain; Uterine Neoplasms
Keywords: Acupuncture; Medicine, Chinese Traditional
MeSH Terms: conditions — Ovarian Neoplasms; Endometriosis; Pelvic Pain; Uterine Neoplasms

INTERVENTIONS:
Procedure: Chinese Acupuncture

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of acupuncture in treating women's health conditions.

DETAILED DESCRIPTION:
This trial comprises three studies. In the first two studies, women will be randomly assigned to receive either real or sham acupuncture therapy. Study 1 will include women with various forms of cancer. White blood cell counts will be used to assess the effects of acupuncture on participants' immune responses. Study 2 will include women with unspecified pelvic pain and endometriosis; a self-report pain scale will be used to assess the effects of acupuncture on participants' symptoms. Study 3 will evaluate the validity and reliability of diagnoses made by Chinese medicine practitioners. In this study, a group of Chinese medicine practitioners will diagnose the same group of patients; consistency of the diagnoses will be evaluated.

ELIGIBILITY:
Inclusion Criteria for Study 1:

* Newly diagnosed ovarian cancer; primary peritoneal cancer; papillary serous cancer of the endometrium; or mixed mesodermal tumor of the uterus, ovary, or fallopian tube
* Currently undergoing chemotherapy
* Meet certain laboratory test requirements

Inclusion Criteria for Study 2:

Currently closed to recruitment

* Diagnosed with endometriosis or unspecified pelvic pain

Exclusion Criteria for Studies 1 and 2:

* Use of white blood cell boosters
* Prior radiotherapy with the exception of whole-breast irradiation for breast cancer
* Prior myelotoxic chemotherapy
* History of symptomatic cardiac or psychiatric disorder
* Use of a pacemaker
* Use of herbs or herbal supplements
* Prior use of acupuncture
* Enrollment in other research studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wayne, PhD, Principal Investigator — New England School of Acupuncture
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States